CLINICAL TRIAL: NCT05961579
Title: A Prospective, Open Label Clinical Study Evaluating the Efficacy and Safety of Cleanser, Serum, and Sunscreen Products for the Treatment of Facial Redness.
Brief Title: Evaluating the Efficacy and Safety of Cleanser, Serum, and Sunscreen Products for Facial Redness.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: RoC Opco LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROC-Rosacea-2023
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Redness
Keywords: facial redness; red
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Intervention Model Description: Subjects will be treated with Barrier Renew Cleanser, Barrier Renew PM Moisturizer, and mineral sunscreen. Cleanser and Barrier Renew PM moisturizer will be used twice daily. Mineral sunscreen will be used every morning and throughout the day as indicated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Barrier Renew Cleanser, Barrier Renew PM Moisturizer, and mineral sunscreen. (Experimental): Enrolled subjects will all receive Barrier Renew Cleanser, Barrier Renew PM Moisturizer, and mineral sunscreen. Cleanser and Barrier Renew PM moisturizer will be used twice daily. Mineral sunscreen will be used every morning and throughout the day as indicated.
  Interventions: Drug: Barrier Renew

INTERVENTIONS:
Drug: Barrier Renew — RoC Skincare (New York, New York, USA) has developed a gentle cleanser and moisturizer that are free of exfoliants, astringents, and other abrasive ingredients. The moisturizer contains emollients, humectants, and silicones to improve the functioning of the skin barrier while antioxidants protect against environmental damage and inflammation

SUMMARY:
The primary objective of this study is to assess the efficacy and safety of combination therapy of a Barrier Renew Cleanser, Barrier Renew PM Moisturizer, and mineral sunscreen in the treatment of redness.

DETAILED DESCRIPTION:
Enrolled subjects will undergo treatment with Barrier Renew Cleanser, Barrier Renew PM Moisturizer, and mineral sunscreen. Cleanser and Barrier Renew PM moisturizer will be used twice daily. Mineral sunscreen will be used every morning and throughout the day as indicated.

Subjects satisfying all inclusion and exclusion criteria will be enrolled in this trial. Prior to receiving any study treatment, mandatory photography using the VISIA system will be done. Patients will return for follow-up assessments at week 2, 4 and 8.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 60 years old (inclusive)
* Subjects must be able and willing to provide written informed consent and photography release
* At the baseline evaluation, all subjects must exhibit all of the following:

  1. Mild to moderate confluent facial redness or blotchy redness
  2. Mild to moderate score (1-6) for tactile roughness or dryness.
* Subject must be in good general health with no other skin disease, disease state or physical condition which would impair evaluation of the areas to be treated or which would increase the subject's health risk by study participation.
* Subjects must have a willingness to minimize sun exposure, avoid direct sun exposure on the face, and avoid the use of tanning beds for the entire duration of the study. Must be willing to wear a hat and reapply sunscreen if sun exposure is unavoidable.
* Subjects must be willing and able to understand and comply with the requirements of the study including minimizing external factors that might trigger redness flare-ups (e.g. spicy foods, excessively hot or cold environments, prolonged sun exposure, strong winds and alcoholic beverages), apply the products as instructed, return for the required treatment period visits, comply with therapy prohibitions, and be able to complete the study.
* For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

  1. A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
  2. Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g., condoms and spermicide), abstinence, and/or vasectomy of partner with a documented second acceptable method of birth control, should the subject become sexually active.

Exclusion Criteria:

* Subjects who are pregnant, planning a pregnancy, or nursing a child.
* Subject using systemic or topical anti-inflammatory agents with the exception of OTC acetaminophen (e.g., Tylenol), ibuprofen (e.g., Advil), or aspirin for 5 days prior to the baseline visit and the duration of the trial
* Subject who could not agree to not use systemic or topical anti-inflammatory agents, with the exception of OTC acetaminophen (e.g., Tylenol), ibuprofen (e.g., Advil), or aspirin during the course of the study.
* Subjects who exhibit severe or advanced redness (persistent deep erythema, telangiectasia forming sprays, papules, pustules, nodules with variable plaque-like edema, or phymatous change).
* Subjects who have used a personal product on the face prior to the study start, which in the opinion of the investigator could interfere with the evaluation of the test articles in the time frame below

  1. Retinoids and other vitamin A derivatives within 1 month
  2. Exfoliating and/or keratolytic products including alpha- or beta-hydroxy acids within 2 weeks
* Subjects who have taken a medication prior to the study start, which in the opinion of the investigator could interfere with the evaluation of the test articles. These medications may include, but are not limited to, the use of any medication to treat rosacea, oral or topical antibiotics, steroids, antifungals, antimicrobials or acne medications for two weeks prior to study start or the time period specified below

  1. Systemic retinoids within 6 months
  2. Systemic tetracycline class antibiotics within 2 months
  3. Systemic macrolide antibiotics within 4 weeks
  4. Initiation of change in hormonal therapy within 3 months
* Subjects with a recent history of atopic dermatitis/eczema or contact dermatitis
* Subjects who are currently under treatment for asthma or diabetes.
* Subjects with any medical condition of the face that could interfere with the study
* Subjects with facial piercings or tattoos that in the Investigator's opinion may hide the diagnosis or disrupt the treatment. Subject agrees not get any facial piercings or tattoos during the study.
* Subjects who are not willing to remove jewelry (earrings), make up and false eyelashes/lash extensions prior to photography.
* Ocular involvement, such as conjunctivitis, episcleritis, iritis, or keratitis.
* History of hypersensitivity or allergy to any of the product ingredients.
* Laser, chemical peel, or surgery on the facial area within 3 months prior to baseline.
* Recent history (<1 year) of substance use disorder
* Subjects that have participated in a clinical research trial in the past 30 days.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-11 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinician Evaluator assessment of change of improvement using the expert grading scale for Redness | Baseline, Day 14, Day 30, Day 60
  Use the following to answer below:
  None= 0 None No erythema or redness of the treatment area
  Mild= 1-3 Mild Slight, but definite redness of the treatment area
  Moderate= 4-6 Moderate Definite redness of the treatment area
  Severe= 7-9 Severe Marked redness of the treatment area
  Using the grading scale above please circle the best answer
  Redness/Erythema= None Mild Moderate Severe
Clinician Evaluator assessment of change of improvement using the expert grading scale for Dryness/Scaling/Roughness | Baseline, Day 14, Day 30, Day 60
  Use the following to answer below:
  None= 0 None No erythema or redness of the treatment area
  Mild= 1-3 Mild Slight, but definite redness of the treatment area
  Moderate= 4-6 Moderate Definite redness of the treatment area
  Severe= 7-9 Severe Marked redness of the treatment area
  Using the grading scale above please circle the best answer
  Dryness/Scaling/Roughness= None Mild Moderate Severe
Clinician Evaluator assessment of change of improvement using the expert grading scale for Luminosity | Baseline, Day 14, Day 30, Day 60
  Use the following to answer below:
  None= 0 None No erythema or redness of the treatment area
  Mild= 1-3 Mild Slight, but definite redness of the treatment area
  Moderate= 4-6 Moderate Definite redness of the treatment area
  Severe= 7-9 Severe Marked redness of the treatment area
  Using the grading scale above please circle the best answer
  Luminosity= None Mild Moderate Severe

SECONDARY OUTCOMES:
Subject Self Assessment Questionnaire | Day 14, Day 30, Day 60
  Agree strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  1. Cleanser/moisturizer helped reduce the redness of my facial skin.
  2. Cleanser/moisturizer calmed and soothed my dry, irritated skin.
  3. Cleanser/moisturizer helped reduce the dryness/tightness of my skin.
  4. Cleanser/moisturizer helped reduce the unevenness of my skin.
  5. Cleanser/moisturizer left my skin radiant/brighter.
  6. Cleanser/moisturizer leaves my skin softer.
  7. Cleanser/moisturizer leaves my skin smoother.
  8. Cleanser/moisturizer soothes my skin.
  9. Cleanser/moisturizer is gentle.
  10. Cleanser/moisturizer makes my skin feel and look less sensitive.
  11. Cleanser/moisturizer regimen leaves skin healthy looking.
  12. Cleanser/moisturizer regimen helped reduce the flakiness of my skin.
  13. Cleanser/moisturizer regimen helped skin to be less reactive.
  14. This simplifies my sensitive skin/rosacea routine.
Clinician Evaluator assessment of change in tolerability Stinging/Burning | Baseline, Day 14, Day 30, Day 60
  Stinging/Burning None (Score of 0) No stinging/burning of the treatment area Mild (Score of 1, 2 or 3) Slight, but definite stinging/burning of the treatment area Moderate (Score of 4, 5 or 6) Definite stinging/burning of the treatment area Severe (Score of 7, 8 or 9) Marked stinging/burning of the treatment area
Clinician Evaluator assessment of change in tolerability Itching | Baseline, Day 14, Day 30, Day 60
  Itching None (Score of 0) No itching of the treatment area. Mild (Score of 1, 2 or 3) Slight, but definite itching of the treatment area. Moderate (Score of 4, 5 or 6) Definite itching of the treatment area that is distracting from daily activities.
  Severe (Score of 7, 8 or 9) Marked itching of the treatment area that wakes you up at night.
Clinician Evaluator assessment of change in tolerability Tightness | Baseline, Day 14, Day 30, Day 60
  Tightness:
  None (Score of 0) No tightness of the treatment area. Mild (Score of 1, 2 or 3) Slight, but definite tightness of the treatment area. Moderate (Score of 4, 5 or 6) Definite tightness of the treatment area. Severe (Score of 7, 8 or 9) Marked tightness of the treatment area.
Clinician Evaluator assessment of change in tolerability Rash | Baseline, Day 14, Day 30, Day 60
  Rash None (Score of 0) No new rash over the treatment area. Mild (Score of 1, 2 or 3) New rash covering some of the treatment area Moderate (Score of 4, 5 or 6) New rash covering much of the treatment area Severe (Score of 7, 8 or 9) New rash covering the entirety of the treatment area

REFERENCES:
- [Background] Schaller M, Almeida LM, Bewley A, Cribier B, Dlova NC, Kautz G, Mannis M, Oon HH, Rajagopalan M, Steinhoff M, Thiboutot D, Troielli P, Webster G, Wu Y, van Zuuren E, Tan J. Rosacea treatment update: recommendations from the global ROSacea COnsensus (ROSCO) panel. Br J Dermatol. 2017 Feb;176(2):465-471. doi: 10.1111/bjd.15173. Epub 2017 Feb 5. PMID 27861741
- [Background] Juliandri J, Wang X, Liu Z, Zhang J, Xu Y, Yuan C. Global rosacea treatment guidelines and expert consensus points: The differences. J Cosmet Dermatol. 2019 Aug;18(4):960-965. doi: 10.1111/jocd.12903. Epub 2019 Feb 26. PMID 30809947
- [Background] Baldwin H, Santoro F, Lachmann N, Teissedre S. A novel moisturizer with high sun protection factor improves cutaneous barrier function and the visible appearance of rosacea-prone skin. J Cosmet Dermatol. 2019 Dec;18(6):1686-1692. doi: 10.1111/jocd.12889. Epub 2019 Feb 25. PMID 30803131